CLINICAL TRIAL: NCT03515187
Title: A Multicenter Randomized Controlled Trial on Prevention and Treatment of Ocular Surface Injury and Meibomian Gland Dysfunction in Patients Using Anti-Glaucoma Eye Drops
Brief Title: Study on Prevention and Treatment of Dry Eye in Patients Using Glaucoma Drops
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Hospital of Southern Medical University (Other)
Responsible Party: Principal Investigator, Yingli Li, Principal Investigator, Shenzhen Hospital of Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LC2016YM017
Record Dates: First submitted 2017-05-13; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Dry Eye; MGD-Meibomian Gland Dysfunction
Keywords: Dug induced dry eye; meibomian gland dysfunction, MGD; Sodium hyaluronate ophthalmic solution; Sodium bromide hydrate eye drops; Meibomian gland massage
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 Medicine treatment group (Experimental): 0.3%sodium hyaluronate ophthalmic solution + 0.1 sodium bromide solution, 28 days
  Interventions: Drug: 0.3% sodium hyaluronate ophthalmic solution; Drug: 0.1% sodium bromide solution
- A2 Combined treatment group (Experimental): 0.3%sodium hyaluronate ophthalmic solution + 0.1 sodium bromide solution，with meibomian gland massage , 28 days
  Interventions: Drug: 0.3% sodium hyaluronate ophthalmic solution; Drug: 0.1% sodium bromide solution; Other: Meibomian gland massage
- B1 Control group (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- B2 Experiment group (Experimental): 0.3%sodium hyaluronate ophthalmic solution, 12 months
  Interventions: Drug: 0.3% sodium hyaluronate ophthalmic solution

INTERVENTIONS:
Drug: 0.3% sodium hyaluronate ophthalmic solution — one to two drops in eye, four times per day
  Arms: A1 Medicine treatment group; A2 Combined treatment group; B2 Experiment group
Drug: 0.1% sodium bromide solution — one to two drops in eye, twice per day
  Arms: A1 Medicine treatment group; A2 Combined treatment group
Other: Meibomian gland massage — Physiotherapy
  Arms: A2 Combined treatment group
Other: Placebo — Vehicle
  Arms: B1 Control group

SUMMARY:
A multicenter randomized controlled trial on prevention and treatment of ocular surface injury and meibomian gland dysfunction in patients using anti-glaucoma eye drops.

DETAILED DESCRIPTION:
1. To compare the efficacy of drug therapy (sodium hyaluronate + sodium bromide) and combined therapy (combined with meibomian gland massage based on drug therapy) on drug-induced dry eye caused by long-term use of anti glaucoma drugs; 2. To evaluate the efficacy of sodium hyaluronate in the prevention of ocular surface and meibomian gland dysfunction and structural damage in the early stage of patients using anti glaucoma eye drops.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age, diagnosed with glaucoma, including primary open-angle glaucoma or primary angle closure glaucoma, require treatment with anti-glaucoma eye drops.
* A group: Patients using glaucoma eye drops longer than 6 months, and in accordance with the diagnostic criteria of dry eye:

  1. Subjective symptoms (required): dryness, foreign body sensation, fatigue and discomfort;
  2. The instability of tear film (required): tear break up time (TBUT);
  3. Lacrimal secretion: Schirmer I test;
  4. The ocular surface damage (strengthen diagnosis): fluorescein staining (FL); in the mentioned in ①+②（TBUT≤5s) or ①+②（TBUT≤10s)+③（<10mm）/④（FL+）。
* The choice of study eyes: Choose the eye of the patient with low basical intraocular pressure, and if the basal intraocular pressure is the same, choose the right eye for the study.
* Voluntary participation in this clinical study, and signed informed consent.

Exclusion Criteria:

* With metabolic diseases, autoimmune diseases, connective tissue diseases, such as diabetes, rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus, Sjogren's syndrome eat;
* Combined with cerebrovascular, liver, kidney, hematopoietic serious system desease, atumor diseases and psychosis.
* Using any artificial tears and except any clinical trials of dry eyes within two weeks.
* With drug therapy, embolization and surgical treatment of dry eyes.
* With other eye diseases, such as eyelid defects, hypophasis, pterygium, chronic dacryocystitis, trichiasis, corneal lesions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Ocular Surface Disease Index (OSDI) score | At screening, 1 month and 2 months for treatment.
  Primary indicator

SECONDARY OUTCOMES:
Change from baseline in Tear break up time (TBUT) | At screening, 1 month and 2 months for treatment.
  Secondary indicator
Change from baseline in corneal staining scores | At screening, 1 month and 2 months for treatment.
  Secondary indicator
Change from baseline in schirmer test | At screening, 1 month and 2 months for treatment.
  Secondary indicator

OTHER OUTCOMES:
Intraocular pressure | At screening, 1 month and 2 months for treatment.
  Additional indicator
Change from baseline in number of blocked meibomian glands | At screening, 1 month and 2 months for treatment.
  Additional indicator

CONTACTS AND LOCATIONS:
Overall Officials: Yingli Li, Study Chair — Shenzhen Hospital of Southern Medicine University; Min Fu, Principal Investigator — Zhejiang Hospital; Lang Bai, Principal Investigator — Nanfang Hospital, Southern Medical University; Guanghua Zhou, Principal Investigator — The Fifth Affiliated Hospital of Southern Medical University; Lei Xi, Principal Investigator — Guangdong Provincial People's Hospital; Xiaolin Zhao, Principal Investigator — Shenzhen Hospital of Southern Medicine University; Wanli Liu, Principal Investigator — Shenzhen Hospital of Southern Medicine University; Yan Wang, Principal Investigator — Shenzhen Hospital of Southern Medicine University; Lina Chen, Principal Investigator — Shenzhen Hospital of Southern Medicine University; Sijing Zhang, Principal Investigator — Shenzhen Hospital of Southern Medicine University; Shingle An, Principal Investigator — Southern Medicine University; Liang Zhang, Principal Investigator — Guangdong Provincial People's Hospital; Ting Meng, Principal Investigator — Zhejiang Hospital
Locations (1):
- Yingli Li, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
If we decided to share the individual participants data (IPD), the IPD will be shared with in six months after the clinical trial by loading ResMan(the web-based medical research public management platform- Research manager, ResMan).